CLINICAL TRIAL: NCT06616220
Title: Dexamethasone for ESPB in Pain Management After Pediatric Idiopathic
Brief Title: Dexamethasone for ESPB in Pain Management After Pediatric Idiopathic Scoliosis Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11/2024
Record Dates: First submitted 2024-09-24; First posted 2024-09-27 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-10

CONDITIONS: Scoliosis; Scoliosis Idiopathic; Scoliosis; Adolescence
MeSH Terms: conditions — Scoliosis | interventions — Dexamethasone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DEXAMETHASONE (Active Comparator): 0.2% ropivacaine + 0.1mg/kg Dexamethasone for erector spinae plane block
  Interventions: Drug: Dexamethasone
- CONTROL (Placebo Comparator): 0.2% ropivacaine for erector spinae plane block
  Interventions: Drug: 0.9%NaCl

INTERVENTIONS:
Drug: Dexamethasone — administration of 0.5ml/kg of 0.2% ropivacaine with 0.1mg/kg Dexamethasone for the erector spine plane block
  Other Names: Dexaethasone
  Arms: DEXAMETHASONE
Drug: 0.9%NaCl — 0.9% NaCl
  Other Names: administration of 0.5ml/kg of 0,2% ropivacaine + 0.01ml/kg 0.9% sodium chloride for the erector spine plane block
  Arms: CONTROL

SUMMARY:
Effect of perineurial dexamethasone on erector spinal plane block duration for pediatric, idiopathic scoliosis surgery.

DETAILED DESCRIPTION:
This study proposes to explore the effect of perineurial Dexamethasone on erector spinal plane block duration for pediatric idiopathic scoliosis surgery.

Children need good analgesia after scoliosis surgery. Peripheral nerve blocks have provided a safe, effective method to control early postoperative pain when symptoms are most severe.

The safety of local anesthesia is essential in children due to the much lower toxicity threshold of local anesthetics. An effective adjuvant, such as Dexamethasone, could allow for a higher dilution of local anesthetics while maintaining and enhancing their analgesic effect.

ELIGIBILITY:
Inclusion Criteria:

* children scheduled for idiopathic scoliosis surgery
* age >10 and <18 years

Exclusion Criteria:

* age < 10 years
* age < 18 years
* infection at the site of the regional blockade
* coagulation disorders
* immunodeficiency
* ASA= or >4
* steroid medication in regular use

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-10-07 (Actual); Study Completion 2025-10-07 (Actual)

PRIMARY OUTCOMES:
First need of opioid analgesia | 48 hours after surgery
  Time after surgery when the patient needs opiate for the first time

SECONDARY OUTCOMES:
Opioid consumption | 48 hours after procedure
  Total opiate consumption after surgery
Numerical Rating Scale [range 0:10] | 4 hours after surgery
  NRS (Numerical Rating Scale; 0 - no pain; 10 - the worst pain ever)
Numerical Rating Scale [range 0:10] | 8 hours after surgery
  NRS (Numerical Rating Scale; 0 - no pain; 10 - the worst pain ever)
Numerical Rating Scale [range 0:10] | 12 hours after surgery
  NRS (Numerical Rating Scale; 0 - no pain; 10 - the worst pain ever)
Numerical Rating Scale [range 0:10] | 24 hours after surgery
  NRS (Numerical Rating Scale; 0 - no pain; 10 - the worst pain ever)
Numerical Rating Scale [range 0:10] | 48 hours after surgery
  NRS (Numerical Rating Scale; 0 - no pain; 10 - the worst pain ever)
Nerve damage [range 0-4] | 12 hours after surgery
  Nerve damage assesment will be performed using the nerve damage score (N0- no nerve damage; N1- minor - sensory paresthesia; N2- major -complete sensory anesthesia; N3- Complete- complete motor defect with or without paraesthesia; N4-CRPS- Complex Regional Pain Syndrome)
Nerve damage [range 0-4] | 24 hours after surgery
  Nerve damage assesment will be performed using the nerve damage score (N0- no nerve damage; N1- minor - sensory paresthesia; N2- major -complete sensory anesthesia; N3- Complete- complete motor defect with or without paraesthesia; N4-CRPS- Complex Regional Pain Syndrome)
Nerve damage [range 0-4] | 48 hours after surgery
  Nerve damage assesment will be performed using the nerve damage score (N0- no nerve damage; N1- minor - sensory paresthesia; N2- major -complete sensory anesthesia; N3- Complete- complete motor defect with or without paraesthesia; N4-CRPS- Complex Regional Pain Syndrome)
glucose | 12 hours after surgery
  blood glucose level
glucose | 24 hours after surgery
  blood glucose level
glucose | 48 hours after surgery
  blood glucose level
MEP | durring surgery
  Motor-Evoced-Potentials

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Spine Diseases and Pediatric Orthopedics, University of Medical Sciences, Poznań, Poland, Poznan, Wielkopolska, Poland

IPD SHARING:
Plan to Share IPD: Yes